CLINICAL TRIAL: NCT01502969
Title: A Phase 2b Study of Rotavin-M1 Vaccine in Vietnamese Children
Brief Title: Safety and Immunogenicity Assessment of Rotavin-M1 in Vietnamese Children
Acronym: Rotavin-M1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Principal Investigator, Dang Duc Anh, Deputy Director, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Rotavin-M1-2b
Record Dates: First submitted 2011-10-29; First posted 2012-01-02 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Diarrhea; Fever; Nausea; Vomit; Irritability
Keywords: diarrhea; fever; nausea; vomit; irritability
MeSH Terms: conditions — Diarrhea; Fever; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Children receiving placebo (cell culture medium in absence of virus)
  Interventions: Biological: cell culture medium in absence of virus
- Rotavirus vaccine (Active Comparator): Rotavin-M1, 10e6.3ffu/dose, 2 doses
  Interventions: Biological: Rotavin-M1

INTERVENTIONS:
Biological: Rotavin-M1 — liquid, 10e6ffu/dose, 2 doses, 2 month interval
  Other Names: KH0118; POLYVAC; G1P[8]
  Arms: Rotavirus vaccine
Biological: cell culture medium in absence of virus — Placebo
  Arms: Placebo

SUMMARY:
This is a multiple-site phase 2b, randomized, placebo control study to evaluate the safety and immunogenicity of Rotavin-M1, produced by the Center for Research and Production of Vaccines and Biologicals, Vietnam.

DETAILED DESCRIPTION:
The investigators evaluate the vaccine schedule consisting of 2 doses of Rotavin-M1, 10e6.3ffu/dose at 2 month interval in children in two study sites, Thanh Son- Phu Tho and Thai Binh city-Thai Binh provinces.

This vaccine dose and schedule was chosen based on results from the previous dose-escalating study (NCT01377571).

ELIGIBILITY:
Inclusion Criteria:

At study entry

1. A healthy male or female, 6 to 12 weeks of age (42 days to 84 days of age).
2. Full term gestation (>=37 weeks).
3. Birth weight of the subject should be >=2.5 kg.
4. Healthy subjects as established by medical history and clinical examination before entering into the study.
5. Did not use any dose of Rota virus vaccine.
6. Written informed consent obtained from the parent or guardian of the subject.

At dose 2

1. Received dose 1.
2. Oral informed consent obtained from the parent or guardian of the subject for continuing participate the study.

Exclusion Criteria:

At study entry

1. Has a chronic disease (cardiovascular, liver, kidney disease).
2. Acute disease at the time of enrolment.
3. Administering corticosteroids (> 1mg/kg/day).
4. Received any immunosuppressive therapy within 4 week before vaccination (Administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
5. Immunosuppressive or immunodeficient condition.
6. Family has immunosuppressive or immunodeficient condition medical history.
7. History of high fever convulsion.
8. Allergic or reaction with any component of vaccine, includes anaphylactic shock with any antibiotic.
9. Preterm of gestation delivery (gestation period < 37 weeks).
10. Low birth weight (<2.5 kg).
11. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
12. Malnutrition.
13. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
14. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.

At dose 2

1. Acute disease at the time of 2nd dose.
2. Administering corticosteroids (> 1mg/kg/day).
3. Received any immunosuppressive therapy within 4 week before vaccination (Administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
4. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
5. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
6. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
7. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 799 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Anti-rotavirus IgA antibody responses 1 month after vaccination | 12 months
  To assess IgA antibody responses 1 month after completing 2 doses of Rotavin-M1, 10e6.3ffu/dose

SECONDARY OUTCOMES:
RV-IgA antibody responses to Rotavin-M1 one year after 1st dose | 12 year
  to assess RV-IgA antibody responses 9 months after the last dose (i.e. 12 months after the 1st dose)
Anti-rotavirus IgG antibody responses 1 month after vaccination with Rotavin-M1 | 12 months
  to assess the anti-rotavirus IgG responses 1 month after completing 2 doses of Rotavin-M1
safety and reactogenicity of each doses of Rotavin-M1, 10e6.3ffu/dose | 12 months
  to assess immediate reations (30 minutes) after administration of each dose of vaccine compared to placebo . To assess adverse events 30 days after each dose of vaccine and placebo, and serious adverse events 1 year after the 1st dose of vaccine and placebo
anti-RV IgG antibody responses 1 year after the 1st dose | 12 month
  To assess anti-RV IgG antibody responses 1 year after the 1st dose of Rotavin-M1 (9 months after the 2nd dose)

CONTACTS AND LOCATIONS:
Overall Officials: Dang D Anh, PhD, Principal Investigator — The National Institute of Hygiene and Epidemiology
Locations (2):
- Vietnam (2):
  - Preventive Medicine Center, Thanh Sơn, Phu Tho
  - Thai Binh Preventive Medicine Center, Thái Bình, Thai Binh

REFERENCES:
- [Background] Anh DD, Thiem VD, Fischer TK, Canh DG, Minh TT, Tho le H, Van Man N, Luan le T, Kilgore P, von Seidlein L, Glass RI. The burden of rotavirus diarrhea in Khanh Hoa Province, Vietnam: baseline assessment for a rotavirus vaccine trial. Pediatr Infect Dis J. 2006 Jan;25(1):37-40. doi: 10.1097/01.inf.0000195635.05186.52. PMID 16395100
- [Background] Nguyen TA, Yagyu F, Okame M, Phan TG, Trinh QD, Yan H, Hoang KT, Cao AT, Le Hoang P, Okitsu S, Ushijima H. Diversity of viruses associated with acute gastroenteritis in children hospitalized with diarrhea in Ho Chi Minh City, Vietnam. J Med Virol. 2007 May;79(5):582-90. doi: 10.1002/jmv.20857. PMID 17385670
- [Background] Ngo TC, Nguyen BM, Dang DA, Nguyen HT, Nguyen TT, Tran VN, Vu TT, Ogino M, Alam MM, Nakagomi T, Nakagomi O, Yamashiro T. Molecular epidemiology of rotavirus diarrhoea among children in Haiphong, Vietnam: the emergence of G3 rotavirus. Vaccine. 2009 Nov 20;27 Suppl 5:F75-80. doi: 10.1016/j.vaccine.2009.08.074. PMID 19931725
- [Background] Van Man N, Luan le T, Trach DD, Thanh NT, Van Tu P, Long NT, Anh DD, Fischer TK, Ivanoff B, Gentsch JR, Glass RI; Vietnam Rotavirus Surveillance Network. Epidemiological profile and burden of rotavirus diarrhea in Vietnam: 5 years of sentinel hospital surveillance, 1998-2003. J Infect Dis. 2005 Sep 1;192 Suppl 1:S127-32. doi: 10.1086/431501. PMID 16088796
- [Background] Kim SY, Goldie SJ, Salomon JA. Cost-effectiveness of Rotavirus vaccination in Vietnam. BMC Public Health. 2009 Jan 21;9:29. doi: 10.1186/1471-2458-9-29. PMID 19159483
- [Background] Luan le T, Trang NV, Phuong NM, Nguyen HT, Ngo HT, Nguyen HT, Tran HB, Dang HN, Dang AD, Gentsch JR, Wang Y, Esona MD, Glass RI, Steele AD, Kilgore PE, Nguyen MV, Jiang B, Nguyen HD. Development and characterization of candidate rotavirus vaccine strains derived from children with diarrhoea in Vietnam. Vaccine. 2009 Nov 20;27 Suppl 5:F130-8. doi: 10.1016/j.vaccine.2009.08.086. PMID 19931712